CLINICAL TRIAL: NCT05718674
Title: Photopheresis in GvHD After Hematopoietic Transplantation: Characteristics of the Procedure and of the Cell Product
Acronym: 3594
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Piccirillo Nicola, Therapeutic Apheresis Director, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3594
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Graft Vs Host Disease; Extracorporeal Photopheresis
Keywords: Extracorporeal Photopheresis
MeSH Terms: conditions — Graft vs Host Disease | interventions — Photopheresis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ECP patient: Patients with chronic or acute GvHD after allogeneic haematopoietic stem cell transplantation undergoing extracorporeal photopheresis
  Interventions: Procedure: Extracorporeal Photopheresis

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis — ECP is performed by collecting leucocytes from the patient through leukopheresis and incubating them with 8-MOP and UVA in extracorporeal circulation. The treatment steps are the collection of leucocytes, photoactivation and subsequent reinfusion of the treated cells.
  Other Names: ECP

SUMMARY:
This is an observational study on extracorporeal photopheresis,an established therapy for the treatment of Graft versus Host Disease (GvHD) post allogeneic haemopoietic stem cell transplantation. There are different techniques and devices to perform cell collection procedure, photoactivation and infusion of mononuclear cells.

The investigators will enrol patients undergoing allogeneic transplants and extracorporeal photopheresis in order to understand whether the different ways in which photopheresis is performed affect cell products and clinical response.

DETAILED DESCRIPTION:
The FPG Stem Cell Transplantation Programme has indicated extracorporeal photopheresis as the therapy of choice for the second-line treatment of steroid-resistant GvHD. If efficacy is supported by clear evidence in the literature, less clear are the mechanism of action, the qualitative and quantitative characteristics of the cells responsible for the clinical response, and the impact of procedural and instrumental variables on clinical efficacy. Indeed, there are different techniques and devices to perform cell collection procedure, photoactivation and infusion of mononuclear cells.

The investigators designed a prospective study that aims to collect data on patients, photopheresis procedures and related cellular products. The analysis of the data will allow the investigators to define the qualitative and quantitative characteristics of the cell products, associating them with the different techniques and instruments, and looking for possible associations with clinical response.

The data collected will be able to contribute to the characterisation of the techniques, procedures and the definition of a minimum cell dose to be treated in order to obtain the response. The aim is to define the volume to be processed or the number of procedures to be carried out by analogy with what is now established practice for the collection procedures of other autologous or allogeneic therapeutic cells (stem cells, lymphocytes, granulocytes), laying the foundations for optimising the treatments and resources employed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of GvHD post allogeneic HSC transplantation being treated with photopheresis;
* signing of informed consent (IC) and consent to personal data processing

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is represented by patients affected by chronic or acute GVHD after allogeneic haematopoietic stem cell transplantation treated at the 'Haematology' and 'Laboratory and DH of Haematology' units undergoing photopheretic treatment in Apheresis Unit of the Fondazione Policlinico Universitario Agostino Gemelli (FPG) - IRCCS.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
The cells | 2 years
  Primary endpoints:
  - To evaluate qualitative and quantitative characteristics of white blood cells in patients undergoing photopheresis. Laboratory tests usually performed in patients undergoing allogeneic transplant and Photopheresis (complete white blood cell count, peripheral blood immunophenotype) will be performed in peripheral blood samples taken before treatment and in samples of cell products collected during treatment. The data obtained will be analysed in relation to the different instruments and techniques used.
WBC in cell product | 2 years
  total WBC count x10^9 collected and infused during ECP
Lymphocytes and Monocytes in cell product | 2 years
  total Lymphocytes and Monocytes count x10^9 collected and infused during ECP
ECP Procedure runtime | 2 years
  Total procedure runtime in minutes
peripheral blood immunophenotype | 2 years
  CD4/CD8 ratio in peripheral blood of patients undergoing ECP
The response | 2 years
  Secondary endpoints:
  - To evaluate the association between the qualitative and quantitative characteristics of white blood cells and the clinical response of patients undergoing photopheresis

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli (FPG) - IRCCS., Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Worel N, Lehner E, Fuhrer H, Kalhs P, Rabitsch W, Mitterbauer M, Hopfinger G, Greinix HT. Extracorporeal photopheresis as second-line therapy for patients with acute graft-versus-host disease: does the number of cells treated matter? Transfusion. 2018 Apr;58(4):1045-1053. doi: 10.1111/trf.14506. Epub 2018 Feb 15. PMID 29446444
- [Background] Bueno JL, Alonso R, Gonzalez-Santillana C, Naya D, Romera I, Alarcon A, Aguilar M, Bautista G, Duarte R, Ussetti P, Cabrera JR. A paired trial comparing mononuclear cell collection in two machines for further inactivation through an inline or offline extracorporeal photopheresis procedure. Transfusion. 2019 Jan;59(1):340-346. doi: 10.1111/trf.14975. Epub 2018 Oct 4. PMID 30284302
- [Background] Brosig A, Hahnel V, Orso E, Wolff D, Holler E, Ahrens N. Technical comparison of four different extracorporeal photopheresis systems. Transfusion. 2016 Oct;56(10):2510-2519. doi: 10.1111/trf.13728. Epub 2016 Jul 26. PMID 27456672
- [Background] Piccirillo N, Putzulu R, Massini G, Fiore AG, Chiusolo P, Sica S, Zini G. Mononuclear cell collection for extracorporeal photopheresis: Concentrate characteristics for off-line UV-A irradiation procedure. J Clin Apher. 2018 Jun;33(3):217-221. doi: 10.1002/jca.21574. Epub 2017 Aug 22. PMID 28833438
- [Background] Piccirillo N, Putzulu R, Massini G, Di Giovanni A, Chiusolo P, Sica S, Zini G. Inline extracorporeal photopheresis: evaluation of cell collection efficiency. Transfusion. 2019 Dec;59(12):3714-3720. doi: 10.1111/trf.15570. Epub 2019 Nov 4. PMID 31682286